CLINICAL TRIAL: NCT01749839
Title: Pain Relief by Platelet-rich Plasma (PRP) Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Saint Bernard Mission University (Other)
Responsible Party: Sponsor
Other Study IDs: NCRM-SBMU0317
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Sciatica
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Past PRP therapy is not sufficient for some part of patients.In this clinical research, The integrated application of PRP with extracellurar matrix and some type of stem cell technique.

ELIGIBILITY:
Inclusion Criteria:

* Injury by professional sports and non professional sports

Exclusion Criteria:

* Other basic disease holder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Athlete community
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The Changes of Amounts of Pain Killer Consumed for Scheduled Term Before and After PRP treatment. | 1 month